CLINICAL TRIAL: NCT03317834
Title: Clinical, Radiographic and Patient-reported Outcomes Associated With the Use of the Navio™ Robotic-assisted Surgical System in Total Knee Arthroplasty
Brief Title: Navio With Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-NPFS-04
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2023-06

CONDITIONS: Total Knee Arthroplasty; Arthroplasty of Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Study Population: Total Knee Replacement with Navio Surgical Systems
  Interventions: Device: Navio ™ Robotic-assisted Surgical System

INTERVENTIONS:
Device: Navio ™ Robotic-assisted Surgical System — Total Knee Replacement

SUMMARY:
The purpose of this study is to demonstrate superior accuracy with the Navio ™ Robotic-assisted Surgical System in achieving desired post-operative mechanical alignment, compared to TKA procedures using standard instruments. An additional study purpose is to document clinical and patient-reported outcomes in subjects receiving TKA with the Navio ™ system.

DETAILED DESCRIPTION:
Total Knee Arthroplasty (TKA) has become an effective and reliable treatment for arthritis of the knee (1). TKA is associated with low morbidity and mortality, and its effectiveness in reducing joint pain and improving range of motion is well established. In 2014, over 750,000 knee replacements were performed in the US (2).

A significant innovation in TKA has been the introduction of computer navigation and robotic-assisted surgery (3). One such technology is the Navio™ Robotic-assisted Surgical System. This system is a semi-autonomous image-free system. During the surgery, the surgeon maps the condylar landmarks and determines alignment indices to define the volume and orientation of bone to be removed. The tools to remove the bone and place the implants are controlled and manipulated by the surgeon with the guidance of a 3-dimensional digital map of the surgical surface.

Originally the Navio™ system was launched for use in unicondylar knee replacement only. To date, there have been over 1000 unicondylar knee replacement surgeries using the system. In 2017, Smith & Nephew Inc. expanded the indications for the Navio™ system to include TKA. The purpose of this multicenter, prospective study is to evaluate outcomes associated with this new indication.

ELIGIBILITY:
Inclusion Criteria:

1. Subject requires primary total knee arthroplasty with the Journey II BCS or Cruciate-Retraining (CR) Systems due to degenerative joint disease (primary diagnosis of osteoarthritis, post-traumatic arthritis, avascular necrosis, rheumatoid arthritis.
2. Subject was considered skeletally mature at the time of cone implantation (at least 18 years or older.)
3. Subject agrees to consent to and to follow the study visit schedule (as defined in the study protocol and informed consent form) by signing the IRB/EC approved informed consent form.
4. Subject plans to be available through two (2) years postoperative follow-up.

Exclusion Criteria:

1. Subject has BMI ≥ 40.
2. Subject has condition(s) that may interfere with the TKA survival or outcome (i.e., Paget's or Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease, or an active, local infection).
3. Subject is deemed by investigator to require a constrained or deep dish tibial insert.
4. Subject has inadequate bone stock to support the device (severe osteopenia, history of severe osteoporosis or severe osteopenia).
5. Subject has mental or neurologic condition(s) that may pre-empt the ability or willingness to restrict activities.
6. Subject is 80 years of age or older.
7. Subject is a prisoner or impending incarceration.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: To eliminate the potential for selection bias, Investigators should screen all subjects undergoing a Navio™ assisted TKA. In order to do so, only the existing information obtained per standard routine medical procedures will be used. No study-specific screening procedures, activities or questionnaires will be performed during pre-screening.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2021-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Lankiewicz, Study Chair — Smith & Nephew, Inc.
Locations (6):
- United States (6):
  - Hedley Orthopedics, Phoenix, Arizona
  - Orthopaedic Associates of Central Arizona, Scottsdale, Arizona
  - San Diego Orthopaedic, San Diego, California
  - Bronson Health, Kalamazoo, Michigan
  - Hospital for Joint Disease Orthopaedic Institute, New York, New York
  - OrthoNeuro, Albany, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment for this study was conducted between 13 November 2017 and 27 May 2021 across six investigative sites.
Period: Overall Study
Arm/Group | Study Population
Started | 122
Completed | 89
Not Completed | 33
Not completed — Death | 2
Not completed — Device Revision | 5
Not completed — Withdrawal by Subject | 13
Not completed — Lost to Follow-up | 13

BASELINE CHARACTERISTICS:
Arm/Group | Study Population
Number analyzed (Participants) | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.51 (8.683)
Age, Customized [Count of Participants; unit: Participants]
  Age Category: < 60 years | 13
  Age Category: >=60 years | 109
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 7
  Race: Other | 8
  Race: White | 107
Region of Enrollment [Number; unit: participants]
  United States | 122
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.32 (5.102)

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With Post-operative Mechanical Alignment
Description: The number of participants achieving post-operative mechanical alignment within ±3 degrees from target with "Yes" indicating mechanical alignment was achieved and "No" indicating mechanical alignment was not achieved.
Time Frame: 1 month
Population: Number of Participants Analyzed indicates the data available for the time frame specified.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Population
Number analyzed (Participants) | 115
Participants
  Yes | 106
  No | 9

2. Secondary Outcome: Count of Participants With Implant Survival
Description: Number of participants with implant survivorship where "No" indicates a revision surgery was not required and "Yes" indicates a revision surgery was required by the 2 year postoperative visit.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Study Population
Number analyzed (Participants) | 122
Participants
  No | 117
  Yes | 5

3. Secondary Outcome: Knee Society Score 2011
Description: The Functional Knee Score is derived from assessments of walking and standing, standard activities, advanced activities, and discretionary activities in Total Knee Arthroplasty (TKA) participants. The 2011 Knee Society Score consists of 4 separate subscales with a higher number indicating a better outcome:
  * A Patient Expectation Score (5items: 15 points, range 0-15)
  * A Functional Activity Score (19 items: 100 points, range 0-100)
  * An "Objective" Knee Score (7 items: 100 points, range 0-100)
  * A Patient Satisfaction Score (5 items: 40 points, range 0-40)
Time Frame: Baseline, 1 month, 6 months, 1 year, and 2 years
Population: Number of Participants Analyzed indicates the data available for the time frame specified.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Population
Number analyzed (Participants) | 122
score on a scale
  Patient Expectation: Baseline | 14.21 (1.627)
  Patient Expectation: 1 Month: number analyzed (Participants) | 114
  Patient Expectation: 1 Month | 8.42 (2.819)
  Patient Expectation: 6 Months: number analyzed (Participants) | 108
  Patient Expectation: 6 Months | 9.78 (3.391)
  Patient Expectation: 1 Year: number analyzed (Participants) | 93
  Patient Expectation: 1 Year | 9.39 (3.040)
  Patient Expectation: 2 Years: number analyzed (Participants) | 87
  Patient Expectation: 2 Years | 9.97 (2.485)
  Functional Activity: Baseline: number analyzed (Participants) | 121
  Functional Activity: Baseline | 42.13 (15.914)
  Functional Activity: 1 Month: number analyzed (Participants) | 112
  Functional Activity: 1 Month | 46.55 (16.155)
  Functional Activity: 6 Months: number analyzed (Participants) | 104
  Functional Activity: 6 Months | 72.28 (15.819)
  Functional Activity: 1 Year: number analyzed (Participants) | 88
  Functional Activity: 1 Year | 79.35 (15.775)
  Functional Activity: 2 Years: number analyzed (Participants) | 83
  Functional Activity: 2 Years | 83.42 (14.931)
  Objective: Baseline: number analyzed (Participants) | 111
  Objective: Baseline | 49.40 (21.382)
  Objective: 1 Month: number analyzed (Participants) | 108
  Objective: 1 Month | 63.02 (17.250)
  Objective: 6 Months: number analyzed (Participants) | 107
  Objective: 6 Months | 78.98 (15.867)
  Objective: 1 Year: number analyzed (Participants) | 90
  Objective: 1 Year | 82.10 (14.339)
  Objective: 2 Years: number analyzed (Participants) | 88
  Objective: 2 Years | 84.51 (13.463)
  Patient Satisfaction: Baseline | 10.93 (6.310)
  Patient Satisfaction: 1 Month: number analyzed (Participants) | 115
  Patient Satisfaction: 1 Month | 22.64 (7.028)
  Patient Satisfaction: 6 Months: number analyzed (Participants) | 109
  Patient Satisfaction: 6 Months | 29.42 (8.358)
  Patient Satisfaction: 1 Year: number analyzed (Participants) | 93
  Patient Satisfaction: 1 Year | 32.19 (7.110)
  Patient Satisfaction: 2 Years: number analyzed (Participants) | 89
  Patient Satisfaction: 2 Years | 33.42 (5.941)

4. Secondary Outcome: Quality of Life EQ-5D-5L
Description: Patient Reported Outcomes using EuroQol Five Dimensions Questionnaire (EQ-5D-5L) was graded on a scale of 0 to 100, with 100 being the best health you can imagine and 0 indicating the worst.
Time Frame: Baseline, 1 Month, 6 Months, 1 Year, 2 Years
Population: Number of Participants Analyzed indicates the data available for the time frame specified.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Population
Number analyzed (Participants) | 122
score on a scale
  Baseline | 73.44 (16.643)
  1 Month: number analyzed (Participants) | 115
  1 Month | 75.01 (12.251)
  6 Months: number analyzed (Participants) | 108
  6 Months | 78.44 (13.462)
  1 Year: number analyzed (Participants) | 93
  1 Year | 81.82 (10.012)
  2 Years: number analyzed (Participants) | 88
  2 Years | 84.18 (9.364)

5. Secondary Outcome: Forgotten Joint Score (FJS)
Description: Forgotten Joint Score (FJS) is a patient-reported outcome measure intended to determine a patient's ability to "forget" about their affected joint after surgery or treatment. The Forgotten Joint Score consists of 12 questions and is scored on a 0-100 scale. The higher the score, the less the patient is aware of their affected joint when performing daily activities.
Time Frame: Baseline, 1 month, 6 months, 1 year, 2 years
Population: Number of Participants Analyzed indicates the data available for the time frame specified.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Population
Number analyzed (Participants) | 122
score on a scale
  Baseline | 11.84 (12.084)
  1 Month: number analyzed (Participants) | 115
  1 Month | 17.31 (19.603)
  6 Months: number analyzed (Participants) | 109
  6 Months | 51.45 (25.377)
  1 Year: number analyzed (Participants) | 93
  1 Year | 66.31 (26.598)
  2 Years: number analyzed (Participants) | 87
  2 Years | 78.56 (26.095)

6. Secondary Outcome: Hospital Length of Stay
Description: Hospital length of stay measured in days
Time Frame: During hospitalization, up to 6 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Study Population
Number analyzed (Participants) | 122
days | 2.04 (0.837)

7. Secondary Outcome: Operative Time
Description: Operative time taken for the surgery measured in minutes.
Time Frame: During surgery, up to 235 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Study Population
Number analyzed (Participants) | 122
minutes | 90.48 (29.316)

8. Secondary Outcome: Radiographic Assessment - Anteroposterior (AP) Angle
Description: AP Angle mechanical alignment of femoral flexion, tibial angle, and total valgus angle
Time Frame: Baseline, 1 month, 6 months, 1 year, and 2 years
Population: Number of Participants Analyzed indicates the data available for the time frame specified.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Study Population
Number analyzed (Participants) | 115
degrees
  Femoral Flexion: Baseline: number analyzed (Participants) | 95
  Femoral Flexion: Baseline | 65.39 (40.711)
  Femoral Flexion: 1 Month | 71.77 (37.265)
  Femoral Flexion: 6 Months: number analyzed (Participants) | 107
  Femoral Flexion: 6 Months | 70.10 (38.357)
  Femoral Flexion: 1 Year: number analyzed (Participants) | 93
  Femoral Flexion: 1 Year | 73.41 (35.754)
  Femoral Flexion: 2 Years: number analyzed (Participants) | 87
  Femoral Flexion: 2 Years | 72.89 (36.198)
  Tibial Angle: Baseline: number analyzed (Participants) | 94
  Tibial Angle: Baseline | 62.34 (38.578)
  Tibial Angle: 1 Month | 69.07 (37.639)
  Tibial Angle: 6 Months: number analyzed (Participants) | 107
  Tibial Angle: 6 Months | 66.59 (38.915)
  Tibial Angle: 1 Year: number analyzed (Participants) | 93
  Tibial Angle: 1 Year | 70.51 (36.435)
  Tibial Angle: 2 Years: number analyzed (Participants) | 87
  Tibial Angle: 2 Years | 70.16 (36.760)
  Total Valgus Angle: Baseline: number analyzed (Participants) | 94
  Total Valgus Angle: Baseline | 126.46 (79.078)
  Total Valgus Angle: 1 Month | 140.15 (74.310)
  Total Valgus Angle: 6 Months: number analyzed (Participants) | 107
  Total Valgus Angle: 6 Months | 136.63 (77.309)
  Total Valgus Angle: 1 Year: number analyzed (Participants) | 93
  Total Valgus Angle: 1 Year | 143.89 (71.527)
  Total Valgus Angle: 2 Years: number analyzed (Participants) | 87
  Total Valgus Angle: 2 Years | 143.05 (72.249)

9. Secondary Outcome: Radiographic Assessment - Lateral Angle
Description: Lateral Angle mechanical alignment of femoral flexion and tibial angle.
Time Frame: Baseline, 1 month, 6 months, 1 year, and 2 years
Population: Number of Participants Analyzed indicates the data available for the time frame specified.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Study Population
Number analyzed (Participants) | 107
degrees
  Lateral Angle Femoral Flexion: Baseline: number analyzed (Participants) | 17
  Lateral Angle Femoral Flexion: Baseline | 6.12 (2.233)
  Lateral Angle Femoral Flexion: 1 Month: number analyzed (Participants) | 105
  Lateral Angle Femoral Flexion: 1 Month | 2.68 (2.600)
  Lateral Angle Femoral Flexion: 6 Months | 2.41 (2.499)
  Lateral Angle Femoral Flexion: 1 Year: number analyzed (Participants) | 93
  Lateral Angle Femoral Flexion: 1 Year | 3.10 (9.465)
  Lateral Angle Femoral Flexion: 2 Years: number analyzed (Participants) | 87
  Lateral Angle Femoral Flexion: 2 Years | 3.31 (9.763)
  Tibial Angle: Baseline: number analyzed (Participants) | 17
  Tibial Angle: Baseline | 80.18 (19.654)
  Tibial Angle: 1 Month: number analyzed (Participants) | 105
  Tibial Angle: 1 Month | 66.30 (37.277)
  Tibial Angle: 6 Months | 63.79 (38.965)
  Tibial Angle: 1 Year: number analyzed (Participants) | 93
  Tibial Angle: 1 Year | 66.56 (38.965)
  Tibial Angle: 2 Years: number analyzed (Participants) | 87
  Tibial Angle: 2 Years | 66.84 (37.326)

10. Secondary Outcome: Radiographic Assessment - Count of Participant Displacements
Description: Number of participants with either no displacement or displacement observed at the 6-month follow-up visit.
Time Frame: 6 months
Population: Number of Participants Analyzed indicates the data available for the time frame specified.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Population
Number analyzed (Participants) | 86
Participants
  No Displacement | 62
  Displacement | 24

11. Secondary Outcome: Radiographic Assessment - Displacement Measurement
Description: Degree of displacement measured in millimeters (mm) for participants with displacement observed at the 6-month follow-up visit.
Time Frame: 6 months
Population: Number of Participants that showed displacement with data available for the time frame specified.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Study Population
Number analyzed (Participants) | 22
millimeters | 3.95 (2.663)

ADVERSE EVENTS:
Time Frame: Time of surgery (i.e., device implantation) through end of the study (2 year post-operative follow-up).
Description: The Intent-to-Treat (ITT) population used for safety analyses and included all consented participants enrolled in the study that received Total Knee Replacement with NAVIO ™ Robotic-assisted Surgical System.
Arm/Group | Study Population
All-Cause Mortality (participants affected / at risk) | 2/122
Serious Adverse Events (participants affected / at risk) | 26/122
Other Adverse Events (participants affected / at risk) | 12/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Population (N=122)
Recurrent dislocation, right hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Quadricep tendon rupture (Musculoskeletal and connective tissue disorders) | 1 (1)
Delayed wound healing (Blood and lymphatic system disorders) | 1 (1)
Arthrofibrosis of total knee arthroplasty (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthrofibrosis right knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Instability of internal left knee prosthesis, init. encounter (Musculoskeletal and connective tissue disorders) | 1 (1)
Patellar tendon tear right knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Prostate cancer (reoccurence) (Reproductive system and breast disorders) | 1 (1)
Deceased, unknown cause (Investigations) | 1 (1)
Rt knee effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Ischemic stroke in left MCA region (Cardiac disorders) | 1 (1)
GI bleed (Gastrointestinal disorders) | 1 (1)
Pulmonary atelectasis J98.11 (Skin and subcutaneous tissue disorders) | 1 (1)
Right ankle fracture (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Periprosthetic infection (Blood and lymphatic system disorders) | 1 (1)
Macular Pucker with surgical repair (Eye disorders) | 1 (1)
Cataracts (Eye disorders) | 1 (1)
Right knee pain, lumbar sprain / strain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in left knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Fall causing torn tendon (Musculoskeletal and connective tissue disorders) | 1 (1)
Infection right knee (Blood and lymphatic system disorders) | 1 (1)
Acquired instability, left knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthrofibrosis (R) knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Left stiffness of knee with history of replacement (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthrofibrosis left knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in right knee (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Population (N=122)
Tooth abcess (Gastrointestinal disorders) | 1 (1)
Wound complication due to suture reaction (Blood and lymphatic system disorders) | 1 (1)
Wound dehiscence (Blood and lymphatic system disorders) | 1 (1)
Pain in left knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in right knee, effusion right knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Iliotibial band friction syndrome - left knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Left knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Pain in left hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Right knee pain, lumbar sprain / strain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT03317834/Prot_SAP_000.pdf